CLINICAL TRIAL: NCT06510374
Title: A Phase 3b, Randomized, Controlled Trial of Nadofaragene Firadenovec vs. Observation in Participants With Intermediate Risk Non-Muscle Invasive Bladder Cancer
Brief Title: Trial of Nadofaragene Firadenovec vs. Observation in Participants With Intermediate Risk Non-Muscle Invasive Bladder Cancer
Acronym: ABLE-32
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000423; U1111-1284-0685 (Other: World Health Organization (UTN))
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-10

CONDITIONS: Intermediate Risk Non-Muscle Invasive Bladder Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 Nadofaragene Firadenovec (Experimental): Participants in the nadofaragene firadenovec arm will receive quarterly instillations with nadofaragene firadenovec for 24 months. For these subjects, the disease evaluation visits will occur within 2 weeks prior to the investigation medicinal products instillation visits.
  Interventions: Drug: Nadofaragene Firadenovec
- Arm 2 - Observation (No Intervention): Subjects will be followed based on the surveillance schedule of the AUA/SUO guideline (quarterly) over the 24 months treatment period.
  .

INTERVENTIONS:
Drug: Nadofaragene Firadenovec — Vector-based gene therapy for NMIBC treatment to potentiate durable therapeutic responses by interferon (IFN) alfa-2b (IFN-α2b) amplification.
  Other Names: Adstiladrin
  Arms: Arm 1 Nadofaragene Firadenovec

SUMMARY:
A phase 3b, Randomized, Controlled Trial of Nadofaragene Firadenovec vs. Observation in Participants with Intermediate Risk Non-Muscle Invasive Bladder Cancer (IR NMIBC)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with intermediate risk non-muscle invasive bladder cancer (IR NMIBC) as defined by American Urological Association (AUA)/Society of Urologic Oncology [SUO] Guideline (2020)
* Has undergone adequate transurethral resection of bladder tumor (TURBT; with or without peri-operative chemotherapy) within 60 days prior to randomization:

  * Recurrence within 1 year, low-grade Ta
  * Solitary low-grade Ta >3 cm
  * Low-grade Ta, multifocal
  * Solitary high-grade Ta, ≤3 cm
  * Low-grade T1

    * Restage TURBT may be done at the discretion of the investigator

Exclusion Criteria:

* Current or previous evidence of muscle invasive (muscularis propria) or metastatic disease presented at the screening visit

High risk NMIBC defined as:

* High-grade T1
* Any recurrent, high-grade Ta
* High-grade Ta >3 cm (or multifocal)
* Any carcinoma in situ (CIS)
* Any Bacillus Calmette-Guérin (BCG) failure in high-grade subject
* Any variant histology
* Any prostatic urethral involvement

Low risk NMIBC defined as:

* First occurrence of low-grade solitary Ta ≤3 cm
* Recurrence of low-grade solitary Ta ≤3 cm >12 months from previous occurrence
* Papillary urothelial neoplasm of low malignant potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence Free survival | 24 months
  Recurrence-free survival, defined as the time from the date of randomization to the date of first documented recurrence, progression or death (due to any cause), whichever occurs first during the treatment period.

SECONDARY OUTCOMES:
Adverse Events | up to 24 months
  Frequency and intensity of adverse events will be recorded from the signed informed consent for participation in the trial up to month 24
Recurrence Free Survival at 12 Months | 12 months
  Recurrence free survival at 12 months defined as whether a subject is alive and is documented recurrence and progression-free for up to 12 months
Recurrence Free Survival at 24 Months | 24 Months
  Recurrence free survival at 24 months defined as whether a subject is alive and is documented recurrence and progression-free for up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceutical
Locations (70):
- United States (36):
  - University of South Alabama (USA) Health System - USACM, Mobile, Alabama
  - Urology Associates of Mobile, Mobile, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Urology Associates of Central California, Fresno, California
  - American Institute of Research, Los Angeles, California
  - Urology Center of Southern California, Murrieta, California
  - University of California, Irvine, Orange, California
  - Advent Health, Denver, Colorado
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - Advanced Urology institute - Pinellas, Largo, Florida
  - Sarasota Memorial Healthcare System, Sarasota, Florida
  - Emory University, Atlanta, Georgia
  - Blessing Health System, Quincy, Illinois
  - Wichita Urology Group, Wichita, Kansas
  - University of Kentucky (UK) - Markey Cancer Center, Lexington, Kentucky
  - Mayo Clinic - Rochester Minnesota, Rochester, Minnesota
  - Specialty Clinical Research of St. Louis, St Louis, Missouri
  - Adult and Pediatric Urology P.C., Omaha, Nebraska
  - Atlantic Health, Morristown, New Jersey
  - Albany Medical College, Albany, New York
  - Great Lakes Physician PC d/b/a Western New York Urology Associates, Cheektowaga, New York
  - AccuMed Research Associates, Garden City, New York
  - Northwell Health -The Arthur Smith Institute for Urology, Lake Success, New York
  - Veterans Affairs New York Harbor Healthcare System - Manhattan VA Medical Center, New York, New York
  - Integrated Medical Professionals, PLLC, New York, New York
  - James J. Peters VA Medical Center, The Bronx, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Oregon Health and Science University (Portland), Portland, Oregon
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Keystone Urology Specialists, Lancaster, Pennsylvania
  - University of Pennsylvania - Perelman Center for Advanced Medicine - Penn Urology, Philadelphia, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Clinics of North Texas PLLC (Dallas), Dallas, Texas
  - Houston Methodist Hospital (Houston), Houston, Texas
  - Urology of Virginia, Virginia Beach, Virginia
- Canada (2):
  - Prostate Cancer Centre, Calgary, Alberta
  - G kenneth Jansz Medicine Professional Corporation, Burlington, Ontario
- France (9):
  - CHU Clermont Ferrand - Hopital Gabriel Montpied, Clermont-Ferrand, Auvergne-Rhône-Alpes
  - CHU Toulouse - Hopital Rangueil, Toulouse, Haute-Garonne
  - CHU Nantes - Hotel Dieu, Nantes, Nantes
  - CHU de Rouen - Hopital Charles-Nicolle, Rouen, Normandy
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux, Nouvelle-Aquitaine
  - Centre Hospitalier Universitaire De Nimes (Nîmes), Nîmes, Occitanie
  - Hospices Civils de Lyon - Edouard Herriot Hosp., Lyon, Rhône-Alps
  - Hopital La Pitie Salpetriere, Paris
  - APHP - Hopital Bichat, Paris, Île-de-France Region
- Japan (15):
  - Aichi Medical University Hospital, Nagakute, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Japanese Red Cross Narita Hospital, Narita, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Hitachi General Hospital, Hitachi, Ibaraki
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - St. Marianna University Hospital, Kawasaki, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Kochi Medical School Hospital, Nankoku, Kochi
  - Mie University Hospital, Tsu, Mie-ken
  - Nara Medical University Hospital, Kashihara, Nara
  - Institute of Science Tokyo Hospital, Bunkyō-Ku, Tokyo
  - Wakayama Medical University Hospital, Wakayama, Wakayama
- Samsung Medical Center, Seoul, Seoul, South Korea
- Spain (7):
  - Instituto de Investigacion Valdecilla (IDIVAL) / Hospital universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Universitario Reina Sofia, Córdoba, Córdoba
  - Hospital Universitario de A Coruna, A Coruña, Galicia
  - Hospital Universitario Virgen De Las Nieves, Granada, Granada
  - Hospital Universitario Basurto, Bilbao, Vizcaya
  - Hospital Universitario 12 De Octubre (Madrid), Madrid

IPD SHARING:
Plan to Share IPD: No